CLINICAL TRIAL: NCT06811558
Title: A Multicenter Head-to-head Comparison of Ixekizumab Vs. Secukizumab in Over 70-year-old Patients with Moderate-to-severe Plaque Psoriasis
Brief Title: Ixekizumab Versus Secukizumab in Over 70-year-old Patients with Psoriasis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024-0283
Record Dates: First submitted 2024-11-18; First posted 2025-02-06 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2024-10

CONDITIONS: Over 70-year-old Patients with Psoriasis
MeSH Terms: interventions — ixekizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ixe. group (Active Comparator)
  Interventions: Biological: Ixekizumab
- Sec. group (Active Comparator)
  Interventions: Biological: Secukizumab

INTERVENTIONS:
Biological: Ixekizumab — injected with ixekizumab
  Arms: Ixe. group
Biological: Secukizumab — injected with secukizumab
  Arms: Sec. group

SUMMARY:
Currently, the main systemic drug therapies in China include methotrexate (MTX), cyclosporine A, retinoids, and biologics. In recent years, monoclonal antibody biologics targeting cellular inflammatory factors have been used in the treatment of severe psoriasis, which is poorly treated with conventional systemic medications, severely affects the quality of life, and is accompanied by significant arthritic symptoms, including tumor necrosis factor-alpha (TNF-alpha) antagonists (etanercept, infliximab, adalimumab); IL-12/23 antagonists (ursodiol, ibuprofen); and IL-12/23 antagonists (ubuntu, ubiquinone). IL-12/23 antagonists (ustekinumab) and IL-17A antagonists (skutecimab). Among them, ezekizumab and stuccizumab are more widely used at present. However, the efficacy, safety, and tolerability of ezekizumab and stuclizumab in the treatment of plaque psoriasis in elderly patients over 70 years of age are not known.

Primary objective:

To evaluate the efficacy of ezekizumab versus secukizumab in patients over 70 years of age with plaque psoriasis.

Secondary objectives:

1. To assess the safety of ezekizumab versus secukizumab in the treatment of patients over 70 years of age with plaque psoriasis;
2. To evaluate the tolerability of ezekizumab versus secukizumab in patients over 70 years of age with plaque psoriasis

DETAILED DESCRIPTION:
Currently, the main systemic drug therapies in China include methotrexate (MTX), cyclosporine A, retinoids, and biologics. In recent years, monoclonal antibody biologics targeting cellular inflammatory factors have been used in the treatment of severe psoriasis, which is poorly treated with conventional systemic medications, severely affects the quality of life, and is accompanied by significant arthritic symptoms, including tumor necrosis factor-alpha (TNF-alpha) antagonists (etanercept, infliximab, adalimumab); IL-12/23 antagonists (ursodiol, ibuprofen); and IL-12/23 antagonists (ubuntu, ubiquinone). IL-12/23 antagonists (ustekinumab) and IL-17A antagonists (skutecimab). Among them, ezekizumab and stuccizumab are more widely used at present. However, the efficacy, safety, and tolerability of ezekizumab and stuclizumab in the treatment of plaque psoriasis in elderly patients over 70 years of age are not known.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women aged ≥70 years; and
2. Diagnosis of plaque psoriasis ≥6 months with or without psoriatic arthritis; and
3. Plaque psoriasis involving ≥3% of body surface area (BSA) at screening and baseline,/Psoriasis Disease Area and Severity Index (PASI) score ≥3, / Static Physician Overall Score (sPGA) ≥ 2 points / DLQI >= 6
4. the subject is suitable for biologic and/or systemic therapy for psoriasis; and
5. The purpose of the trial is well understood, and the pharmacological effects and possible adverse reactions of the test drug are well understood; the subject will be treated according to Hull's guidelines.
6. The subject has a basic understanding of the purpose of the trial, the pharmacological effects of the test drug and the possible adverse effects; and (6) The subject has voluntarily signed an informed consent form in the spirit of the Declaration of Helsinki.

Exclusion Criteria:

1. With other severe skin diseases, tumors, other systemic diseases (e.g., inflammatory bowel disease), or psychiatric disorders;
2. With tuberculosis, HIV, hepatitis B, hepatitis C and other infections;
3. Those who are allergic to ezekizumab or stavudine;
4. Those who have received other systemic therapies (including but not limited to glucocorticoids, cyclosporine, methotrexate, avitamin A, azathioprine, hydroxychloroquine, thalidomide, etc.) within the previous 4 weeks;
5. Those who have participated in other clinical trials in the previous 3 months;

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects who improved their PASI score by 90% (PASI 90) or more from baseline or achieved an sPGA score of 0 or 1 at Week 16. | Week 16

SECONDARY OUTCOMES:
Proportion of subjects with 100% improvement in PASI score from baseline at Week 16 | Week 16
At Week 16, the proportion of subjects with an sPGA score of 0 | Week 16
Absolute value of change from baseline in subjects' PASI, sPGA, BSA, DLQI, and NRS at Week 16 | Week 16
atients who achieved a PASI of 90 at week 16. | Week 16
patients who achieved PASI 75 at week 16 | Week 16

IPD SHARING:
Plan to Share IPD: No